CLINICAL TRIAL: NCT04207255
Title: A Phase II Study of the Addition of Opaganib to Androgen Antagonists in Patients With Prostate Cancer Progression on Enzalutamide or Abiraterone
Brief Title: Addition of Opaganib to Androgen Antagonists in Patients With mCRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00095537; 1P01CA203628-01 (NIH); 103193 (Other: MUSC)
Record Dates: First submitted 2019-11-25; First posted 2019-12-20 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: Yeliva; ABC294640; 103193
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide; abiraterone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 2: Opaganib with abiraterone (Experimental)
  Interventions: Drug: Opaganib; Drug: Abiraterone
- Cohort 3: Opaganib with enzalutamide (Experimental)
  Interventions: Drug: Opaganib; Drug: Enzalutamide
- Cohort 1a: Opaganib with abiraterone (Experimental)
  Interventions: Drug: Abiraterone; Drug: Opaganib
- Cohort 1b: Opaganib with enzalutamide (Experimental)
  Interventions: Drug: Enzalutamide; Drug: Opaganib

INTERVENTIONS:
Drug: Opaganib — 500mg of Opaganib orally twice a day continuously.
  Arms: Cohort 2: Opaganib with abiraterone; Cohort 3: Opaganib with enzalutamide
Drug: Abiraterone — IV as directed by SOC
  Arms: Cohort 1a: Opaganib with abiraterone; Cohort 2: Opaganib with abiraterone
Drug: Enzalutamide — IV as directed by SOC
  Arms: Cohort 1b: Opaganib with enzalutamide; Cohort 3: Opaganib with enzalutamide
Drug: Opaganib — 250mg of Opaganib orally twice a day continuously.
  Arms: Cohort 1a: Opaganib with abiraterone; Cohort 1b: Opaganib with enzalutamide

SUMMARY:
This is a Phase II study of the investigational drug opaganib. Patients with metastatic castration resistant prostate cancer (mCRPC) who have experienced disease progression while receiving abiraterone or enzalutamide will receive Opaganib at either 250 mg or 500 mg by mouth twice a day continuously. Patients will continue on study drug until the development of progressive disease, intolerable toxicity, withdrawal of patient consent or other event as outlined in patient discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have mCRPC. Each patient must have:

   * Tissue diagnosis documented by pathology report, or clinic note attesting to same.
   * Radiographically-demonstrated metastases
   * Patients must have adenocarcinoma, or ductal carcinoma, or combinations of these two entities
2. Voluntary, signed and dated, institutional review board (IRB)-approved informed consent form in accordance with regulatory and institutional guidelines.
3. Documented progression during treatment with enzalutamide or abiraterone, as determined by the enrolling investigator.
4. Testosterone level documented to be less than 50ng/
5. 18 years of age or older.
6. ECOG performance status of 0-2.
7. Acceptable liver function:

   * Bilirubin ≤ 1.5 times upper limit of normal (CTCAE Grade 1 baseline)
   * AST (SGOT) & ALT (SGPT) ≤ 3 x ULN (CTCAE Grade 1 baseline)
   * Subjects with Gilbert's syndrome may be included if the total bilirubin is <3x ULN and the direct bilirubin is within normal limits
8. Acceptable kidney function indicated by serum creatinine ≤ 1.5 X ULN (CTCAE Grade 1 baseline)
9. Acceptable hematologic status:

   * Absolute neutrophil count ≥ 1000 cells/mm3,
   * Platelet count ≥ 75,000 (plt/mm3) (CTCAE Grade 1 baseline)
   * Hemoglobin ≥ 9.0 g/dL.
10. Fasting blood glucose of <165mg/dL
11. Urinalysis: no clinically significant abnormalities
12. International normalized ratio (INR) ≤1.7
13. Well-controlled blood pressure as determined by the treating investigator
14. Patients requiring narcotic analgesics must be on stable doses for at least 2 weeks prior to study entry.

Exclusion Criteria:

1. New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG.
2. Underlying psychiatric disorder requiring hospitalization within the last two years.
3. Clinically significant neurological disorder (Parkinson's disease, dementia, multiple sclerosis), as determined by the enrolling investigator.
4. Active, uncontrolled bacterial, viral or fungal infection, requiring systemic therapy.
5. Treatment with radiation therapy, surgery, or investigational therapy within 28 days prior to registration.
6. Unwillingness or inability to comply with procedures required in this protocol.
7. Serious nonmalignant disease that could compromise protocol objectives in the opinion of the Investigator.
8. Patients who are receiving coumadin, apixaban, argatroban or rivaroxaban. Patients who are receiving other drugs that are sensitive substrates of CYP450 1A2, 3A4, 2C9, 2C19 or 2D6, or strong inhibitors or inducers of all major CYP450 isozymes that cannot be stopped at least 7 days or 5 half-lives (whichever is longer) before starting treatment with opaganib may be treated on this study with careful monitoring for toxic effects or loss of efficacy of the relevant drug. A list of commonly used drugs that are sensitive substrates of CYP450 1A2, 3A4, 2C9, 2C19 or 2D6, or strong inhibitors or inducers of all major CYP450 isozymes with the half-life of each drug identified, is included as an Appendix C.
9. Patients who are currently participating in any other clinical trial of an investigational product.
10. Other primary malignancy requiring systemic treatment within past 5 years except carcinoma in situ of the cervix or urinary bladder or non-melanoma skin cancer.
11. Any other mental incapacitation or psychiatric illness that would preclude study participation, as determined by the enrolling investigator.
12. Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 2: Opaganib With Abiraterone | Cohort 3: Opaganib With Enzalutamide | Cohort 1a: Opaganib With Abiraterone | Cohort 1b: Opaganib With Enzalutamide
Started | 27 | 36 | 3 | 3
Completed | 27 | 36 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 2: Opaganib With Abiraterone | Cohort 3: Opaganib With Enzalutamide | Cohort 1a: Opaganib With Abiraterone | Cohort 1b: Opaganib With Enzalutamide | Total
Number analyzed (Participants) | 27 | 36 | 3 | 3 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 11 | 1 | 0 | 16
  >=65 years | 23 | 25 | 2 | 3 | 53
Age, Continuous [Mean (Full Range); unit: years] | 71 [55 to 87] | 71 [57 to 88] | 67 [65 to 70] | 71 [68 to 73] | 71 [55 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 27 | 36 | 3 | 3 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 25 | 34 | 3 | 3 | 65
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 9 | 0 | 0 | 19
  White | 17 | 26 | 3 | 3 | 49
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Status
Description: Stable disease or better according to Prostate Cancer Working Group 3 (PCWG3) criteria after four cycles of treatment
Time Frame: 113 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Opaganib With Abiraterone | Cohort 3: Opaganib With Enzalutamide | Cohort 1a: Opaganib With Abiraterone | Cohort 1b: Opaganib With Enzalutamide
Number analyzed (Participants) | 27 | 36 | 3 | 3
Participants | 4 | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years, 9 months, 23 days
Arm/Group | Cohort 2: Opaganib With Abiraterone | Cohort 3: Opaganib With Enzalutamide | Cohort 1a: Opaganib With Abiraterone | Cohort 1b: Opaganib With Enzalutamide
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/36 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/27 | 11/36 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 27/27 | 36/36 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2: Opaganib With Abiraterone (N=27) | Cohort 3: Opaganib With Enzalutamide (N=36) | Cohort 1a: Opaganib With Abiraterone (N=3) | Cohort 1b: Opaganib With Enzalutamide (N=3)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular Dysrythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 2: Opaganib With Abiraterone (N=27) | Cohort 3: Opaganib With Enzalutamide (N=36) | Cohort 1a: Opaganib With Abiraterone (N=3) | Cohort 1b: Opaganib With Enzalutamide (N=3)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 1 (1) | 0 (0)
Rigors (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Limb edema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal cramping (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hand pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Leg cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Leg weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized weakness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual disturbances (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral dysethesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
APTT increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Altered mental status (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Belching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disorientation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection at port site (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart palpatations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT04207255/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT04207255/ICF_001.pdf